CLINICAL TRIAL: NCT07052058
Title: Triple-Blind Randomized Clinical Trial of Tocilizumab vs Placebo: Potential Use of an IL-6 Antagonist as an Adjuvant to Standard Treatment for Treatment-Resistant Major Depression in the Brazilian Public Health System (SUS)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-0245; 88904825.7.0000.5327 (Other: Plataforma Brasil)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Treatment-Resistant Major Depressive Disorder
MeSH Terms: interventions — tocilizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tocilizumab (Experimental)
  Interventions: Biological: Tocilizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Normal Saline (0.9% NaCl)
- Healthy controls, for comparison of inflammatory biomarkers (No Intervention): Healthy controls (HCs) will be recruited for comparison of CRP and IL-6 levels. They will be required to have no current or past history of psychiatric disorders as assessed by the SRQ-20, an instrument developed by the WHO to measure the level of suspicion of mental disorders.

INTERVENTIONS:
Biological: Tocilizumab — Single infusion tocilizumab, 8 mg/kg, diluted in 100 mL of normal saline
  Arms: Tocilizumab
Drug: Normal Saline (0.9% NaCl) — Placebo, same volume as intervention
  Arms: Placebo

SUMMARY:
Clinical trial aimed at evaluating whether a single infusion of tocilizumab, a medication that blocks the action of an inflammatory molecule called interleukin-6 (IL-6), can reduce symptoms of treatment-resistant major depression compared to placebo in non-hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Provide informed consent Understand written and spoken Portuguese Able and willing to consent to blood sampling Willing to abstain from strenuous exercise for 72 hours prior to assessment Meet DSM-5/MINI criteria for a diagnosis of depression resistant to at least two adequate courses of treatment at the time of eligibility assessment Serum/plasma hsCRP level ≥3 mg/L

Exclusion Criteria:

Diagnosis of bipolar disorder or personality disorder History of substance use disorder in the past six months. Presence of active infection (TB, Hepatitis B, Hepatitis C or HIV) or autoimmune disease Pregnancy or breastfeeding History of significant cardiovascular disease, recent cancer, or hematological disorders BMI >40 kg/m² or weight >100 kg Hypersensitivity to tocilizumab or any of its excipients. CRP ≥20 mg/L

Inclusion criteria to the 10 healthy controls recruited for comparison of inflammatory biomarkers:

Age ≥ 18 No current or lifetime psychiatric diagnosis, as measured by the SRQ-20 Provide informed consent Understand written and spoken Portuguese Able and willing to consent to blood sampling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2029-07-29 (Estimated); Study Completion 2029-07-29 (Estimated)

PRIMARY OUTCOMES:
Clinical global improvement (CGI) | Baseline and follow-ups (day 7, day 14, day 28 and month 6)
Reduction in depressive symptoms (HDRS) | Baseline and follow-ups (day 7, day 14, day 28 and month 6)
General psychiatric symptoms improvement (BPRS) | Baseline and follow-ups (day 7, day 14, day 28 and month 6)
ECT indication after invervention | Follow-ups (day 7, day 14, day 28 and month 6)

SECONDARY OUTCOMES:
Cognitive performance (Montreal Cognitive Test) | Baseline and follow-ups (day 7, day 14, day 28 and month 6)
Quality of life (EUROHISQOL8) | Baseline and follow-ups (day 7, day 14, day 28 and month 6)
Psychiatric hospitalization rate in 6 months | 6 months follow-up
Suicidal ideation (MINI) | Elegibility and follow-ups (day 7, day 14, day 28 and month 6)
Quality of life (WHOQOL-BREF) | Baseline, follow-ups (day 7, day 14, day 28 and month 6)

CONTACTS AND LOCATIONS:
Overall Officials: Neusa Sica da Rocha, PhD, Study Director — Federal University of Rio Grande do Sul (UFRGS)
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No